CLINICAL TRIAL: NCT06484855
Title: A Double Blind, Randomized Study Assessing the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Doses of IBI355 in Patients With Primary Sjogren's Syndrome
Brief Title: Safety and Tolerability of IBI355 in Patients With Primary Sjogren's Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI355A102
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Primary Sjögren's Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IBI355 7.5mg/kg (Experimental): IBI355 7.5mg/kg and placebo will be given to the subjects every 4 weeks (8:2)
  Interventions: Drug: IBI355; Drug: IBI355 placebo
- IBI355 15mg/kg (Experimental): IBI355 15mg/kg and placebo will be given to the subjects every 4 weeks (8:2)
  Interventions: Drug: IBI355; Drug: IBI355 placebo
- IBI355 30mg/kg (Experimental): IBI355 30mg/kg and placebo will be given to the subjects every 4 weeks (8:2)
  Interventions: Drug: IBI355; Drug: IBI355 placebo

INTERVENTIONS:
Drug: IBI355 — IBI355 IV. Q4W
Drug: IBI355 placebo — IBI355 placebo IV. Q4W

SUMMARY:
This study aims to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple ascending doses of IBI355 in primary Sjogren's syndrome (pSS) patients. This study also aims to evaluate the anti-Drug antibody after multiple ascending doses of IBI355 in pSS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and sign the informed consent form;
2. Age ≥ 18 years, male or female；
3. Body Mass Index (BMI) within the range of 18.0 to 28.0 kg/m² (inclusive);
4. Meet the 2016 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria for Sjögren's Syndrome;
5. Positive for anti-Sjögren's syndrome A autoantibodies (SSA) and/or anti-Sjögren's syndrome B autoantibodies (SSB);
6. Unstimulated whole salivary flow rate > 0 ml/min;

Exclusion Criteria:

1. Individuals who have had allergic reactions to any components of IBI355, have allergic diseases, or possess an allergic constitution;
2. Those who cannot tolerate frequent venipuncture procedures;
3. Participants diagnosed with secondary Sjögren's syndrome, or whose clinical symptoms (or laboratory abnormalities) require explanation by another connective tissue disease (such as systemic lupus erythematosus, mixed connective tissue disease, etc.).
4. Subjects paticipated in the other clinical trail in 1 month or less than 5 t1/2 since the previous clinical trial (which is longer)；
5. Subjects with an infection requiring systemic medication was present within 30 days prior to randomization;
6. HIV-Ab、RPR、HCV-Ab、HBV、HBeAg or HBcAb, one of them positive;
7. There have a clinical or imaging evidence that the subject with active tuberculosis, or there is evidence that the subject is in the incubation period for tuberculosis;

6.Patients with a history of central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, metabolic disorders and other systemic diseases; 7. Subject with a hcg positive; 8.Patients with a history of neuropsychiatry or who are considered unfit to participate in this clinical trial; 9.Patients with pulmonary interstitial fibrosis, or those requiring combined antifibrotic drug therapy, or those with abnormal lung function that the investigators determined was not suitable for this study; 10. Need to use other drugs that could cause xerostomia during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-14 (Actual); Primary Completion 2025-06-21 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events | up to week 24

SECONDARY OUTCOMES:
Area under the Curve(AUC) of multi-dose of IBI355 | Up to week 16
Peak serum concentration(Cmax) of multi-dose of IBI355 | Up to week 16
Clearance (CL) of multi-dose of IBI355 | Up to week 16
Half-life (t1/2) of multi-dose of IBI355 | Up to week 16
The ratio of Anti-drug antibody of multi-dose of IBI355 | Up to week 24

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No